CLINICAL TRIAL: NCT06539780
Title: Imagery Rescripting for Early Psychosis: a Multiple-Baseline Single-Case Experimental Design.
Brief Title: Imagery Rescripting as a Treatment for Early Psychosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Judy Luigjes, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A2023.0217.0001
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Psychosis; Psychotic Disorders; Schizophrenia; Psychoses, Traumatic
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Neurocognitive Disorders

STUDY DESIGN:
Intervention Model Description: Multiple baseline case series design: Patients wil be randomized to different lengths of baseline period and the effectiveness of the treatment is tested by comparing means and slopes of daily reported schema- or core beliefs, wellbeing and self esteem. Also psychotic and trauma symptoms will be measured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imagery Rescripting (Experimental): Baseline consists of a random assigned period of 1-3 weeks with measurements and no intervention.
  Intervention consists of a maximum of 6 sessions of imagery rescripting, provided twice-weekly.
  Post treatment follow up consists of 3 weeks with only measurements and no intervention.
  Interventions: Behavioral: Imagery Rescripting

INTERVENTIONS:
Behavioral: Imagery Rescripting — In Imagery Rescripting participants imagine a different sequence of events based on missed emotional needs and rescript until needs are fulfilled. Duration of sessions is up to 60 minutes.

SUMMARY:
The goal of this multiple baseline case series study is to test the effect of imagery rescripting (ImRs) in early psychosis.

Primary objective :The course of schema or core beliefs, wellbeing and self-esteem in early psychosis.

Secondary objective: The change in psychotic and trauma symptoms (full questionnaire), core emotions, strength of affect and obtrusiveness of image.

Other objectives are research into the working mechanisms of imagery rescripting by collecting qualitative data from patients and their practitioner in a qualitative interview.

For this study, a multiple-baseline single-case experimental design (SCED) is used testing different outcome variables in 8 patients with early psychosis. After a variable baseline period of 1-3 weeks participants will start twice weekly with imagery rescripting for 4-6 sessions, followed by a 3 week follow up.

Participants will rate schema- or core beliefs on a visual analogue scale. Wellbeing and selfesteem will be measured 4 times with questionnaires. In addition . Secondary we will asses four times questionnaires about psychotic and trauma symptoms and daily measures of core emotions, affect and obtrusiveness of the intrusion. After treatment participants will be interviewed about their experiences.

DETAILED DESCRIPTION:
In a multiple baseline case series study the effectiveness of Imagery Rescripting (ImRs) as a treatment for Early Psychosis will be researched. 5-10 participants with a diagnosis of psychosis will be randomized to a waiting list with variable length between 1-3 weeks. After this participants will enter the ImRs (approximately 4-6 sessions), given twice-weekly. Follow up assessment will take place 3 weeks after ending treatment. Primary outcome is schema of core beliefs, wellbeing and self esteem, operationalized by daily measures with visual analogue scales and questionnaires 4 times like the MHQoL and the RSAS. Secondary outcomes are psychotic symptoms (PSYRATS) and trauma symptoms (PCL-5) (measured 4 times), strength of affect and obtrusiveness of image (measured daily with VAS scales).

The hypothesis is that the primary outcomes will reduce more during the intervention phase compared to the baseline phase and remain stable or even further improve in the follow-up phase. For the secondary outcomes the investigator hypothesized a decrease in psychotic and trauma symptoms and less strength of affect and obtrusiveness of image.

The largest effect is expected from pre- to post treatment, with a relative stable little change during baseline and follow-up.

Results will be analyzed using visual inspection, repeated measures ANOVA and multilevel analysis, pooling the effects of the individual cases. Finally, participants will be interviewed post treatment about their experiences during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria for schizophrenia spectrum disorder, a primary diagnosis according to the Diagnostic and Statistical Manual of Mental Disorders (5th ed; American Psychiatric Association, 2013)
* Preferably Dutch literacy, as exception English literacy is allowed if the practitioner is able to provide treatment
* Preferably stable in medication at start.

Exclusion Criteria:

* Current mania
* Active suicidal plans
* Current alcohol or drugs abuse as diagnosed by DSM-5, use is permitted if not significantly influencing treatment outcomes.
* Neurological disorder

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Schema or core beliefs | 7-9 weeks
  Idiosyncratic schema- or core beliefs related to the early psychosis, VAS scales with range 0-100. A higher score indicates symptom severity.
Wellbeing | 4 times: at start, end baseline (up to 3 weeks), after treatment (expected 3 weeks after start of intervention), at follow up (3 weeks after ending treatment)
  The MHQoL measures wellbeing. The minimum score is 1 and the maximum score is 21. A higher score indicates more wellbeing.
Self Esteem | 4 times: at start, end baseline (up to 3 weeks), after treatment (expected 3 weeks after start of intervention), at follow up (3 weeks after ending treatment)
  The Rosenberg Self-Esteem Scale (RSAS) measures self esteem. The minimum score is 0 and the maximum score is 30. A higher score indicates more self esteem.

SECONDARY OUTCOMES:
Psychotic symptoms | 2 times: at start and after ending treatment
  The PSYRATS measures psychotic symptoms. The total score ranges from 2 to 41, with higher scores indicating more severe symptoms. The Psychotic Symptom Rating Scale (PSYRATS) is comprised of 17 items on specific dimensions of hallucinations and delusions, with each item being rated from 0 (absent) to 4 (severe).
Trauma Symptoms | 2 times: at start and after ending treatment
  The PCL-5 measures traumatic symptoms. The PTSD Checklist for DSM-5 is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms. Respondents are asked to rate how bothered they have been by each of 20 items in the past month on a 5- point Likert scale ranging from 0-4. Items are summed to provide a total severity score (range = 0-80).
Strength of affect | 7-9 weeks
  Strength of affect is measured by a visual analogue scale (VAS scale) on a range of 0-100, measured daily, with higher scores indicating more severe symptoms
Obtrusiveness of image | 7-9 weeks
  Obtrusiveness is measured by a visual analogue scale (VAS scale) on a range of 0-100, measured daily, with higher scores indicating more severe symptoms
Emotions | 7-9 weeks
  Idiosyncratic emotions (e.g. shame of guilt) are measured by a visual analogue scale (VAS scale) on a range of 0-100, measured daily, with higher scores indicating more severe symptoms

OTHER OUTCOMES:
Qualitative Interview | Post treatment up to 3 months
  With an interview, participants will be interviewed after treatment. A qualitative analysis will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Damiaan Denys, Prof, Principal Investigator — Amsterdam UMC; Arnoud Arntz, Prof., Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam-Zuidoost, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
No Due to privacy regulations patient data will not be shared unless the European Union (EU) regulations on data protection are guaranteed.